CLINICAL TRIAL: NCT04669691
Title: A Phase 2, Randomized, Observer-Blind, Multicenter Study to Evaluate the Immunogenicity and Safety of Several Doses of Antigen and MF59 Adjuvant Content in a Monovalent H5N1 Pandemic Influenza Vaccine in Healthy Pediatric Subjects 6 Months to < 9 Years of Age
Brief Title: A Dose-ranging Pediatric Study of an Adjuvanted Pandemic Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V87_30; 2016-001898-32 (EudraCT Number)
Record Dates: First submitted 2016-11-30; First posted 2020-12-17 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Influenza, Human
Keywords: Pandemic; Influenza; Vaccine; MF59; Adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lowest dose, less adjuvant aH5N1 vaccine (Experimental): Two consecutive intramuscular (IM) administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant
- Low dose, less adjuvant aH5N1 vaccine (Experimental): Two consecutive IM administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant
- Mid dose, less adjuvant aH5N1 vaccine (Experimental): Two consecutive IM administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant
- Lowest dose, adjuvanted aH5N1 vaccine (Experimental): Two consecutive IM administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant
- Low dose, adjuvanted aH5N1 vaccine (Experimental): Two consecutive IM administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant
- Mid dose, adjuvanted aH5N1 vaccine (Experimental): Two consecutive IM administrations (Day 1 and Day 22)
  Interventions: Biological: H5N1 antigen combined with MF59 adjuvant

INTERVENTIONS:
Biological: H5N1 antigen combined with MF59 adjuvant — Eligible subjects will be stratified by age at the time of enrollment into one of 2 age cohorts and within each age cohort will be randomly assigned (equally) to 1 of 6 study vaccine groups. Subjects in each study vaccine group will be scheduled to receive 2 injections of aH5N1 vaccine 3 weeks apart
  Other Names: aH5N1

SUMMARY:
This study is a pediatric dose-ranging study to evaluate the safety and immunogenicity of vaccination with different MF59-adjuvanted H5N1 vaccine formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects of 6 months through <9 years of age on the day of informed consent/assent.
2. Documented consent provided by the subject's parent(s)/LAR(s) have voluntarily given written informed consent/assent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
3. Subject's parent(s)/LAR(s) able to comprehend and comply with all study procedures, and available for all clinic visits and telephone contacts scheduled in the study.
4. Subjects must provide a baseline blood sample within 10 days prior to the Day 1 vaccination.

Exclusion Criteria:

Each subject must not have:

1. Progressive, unstable or uncontrolled clinical conditions.
2. Hypersensitivity, including allergy, to any component of vaccines, medicinal products or medical equipment whose use is foreseen in this study.
3. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws, ie,

   1. Subjects who have had a fever (body temperature measurement ≥ 38°C) within three days prior to vaccination. The subject may return for vaccination after they have been free of fever for three days.
   2. History of epilepsy or convulsions (excluding febrile convulsions).
   3. A subject who has any medical condition meeting the definition of AESI defined for the purposes of this trial (see appendix A).
   4. Subjects who have received antipyretic medication within the past 24 hours prior to vaccination. The subject may return for vaccination after a period of 24 hours has passed since the administration of an antipyretic.
4. Abnormal function of the immune system resulting from:

   1. Clinical conditions.
   2. Systemic administration of corticosteroids (PO/IV/IM) for more than 14 consecutive days within 90 days prior to informed consent/assent. Topical, inhaled and intranasal corticosteroids are permitted. Intermittent use (one dose in 30 days) of intra-articular corticosteroids are also permitted.
   3. Administration of antineoplastic and immunomodulating agents or radiotherapy from within 90 days prior to informed consent/assent.
5. Suspicion of pandemic influenza illness within past six months or have ever received previous pandemic H5N1 flu vaccination.
6. Received immunoglobulins or any blood products within 180 days prior to informed consent/assent.
7. Received an investigational or non-registered medicinal within 30 days prior to informed consent/assent.
8. Children of study site staff (this includes research or clinic staff) or children who are otherwise related to study site staff or have household members who are study site staff. Study site staff are employees with direct or indirect contact with study subjects and/or have access to any study documents containing subject information. This would include receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians, medical assistants, document scanners, etc. study personnel as an immediate family or household member.
9. Any other clinical condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subject due to participation in the study.
10. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine prior to day 43. Following day 43 other vaccines may be administered, including seasonal flu.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2020-12-19 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Manager, Study Director — Seqirus
Locations (7):
- Estonia (2):
  - 23302- Al Mare Perearstikeskus OÜ, Tallinn, Harju
  - 23301- Clinical Research Center, Tartu, Tartu
- Philippines (5):
  - 60805 - De La Salle Medical and Health Sciences Institute, Dasmariñas, Manila
  - 60804 - University of Perpetual Help Dalta Medical Center, Las Piñas, Manila
  - 60802- Philippine General Hospital, Manila, National Capital Region
  - 60803- Philippine General Hospital - Pediatrics, Manila, National Capital Region
  - 60801- Philippine General Hospital - Pediatrics, Manila

IPD SHARING:
Plan to Share IPD: Yes
SEQIRUS supports the release of anonymized subject-level and study-level data in compliance with regulatory requirements, including Clinical Documents which are part of the CTD modules submitted to regulatory agencies for public release.
  Summary results disclosure is either in document form (e.g., ICH E3 Clinical Study Report synopsis) or structured data form (such as summary results in ClinicalTrials.gov (United States) or eudract.ema.europa.eu (EU Clinical Trial Registry [EU CTR])
Supporting Information: Study Protocol, SAP
Time Frame: SEQIRUS discloses results from clinical studies within 12 months of last patient last visit (LPLV) unless otherwise mandated by local laws or regulations.
Access Criteria: SEQIRUS will consider requests from qualified scientific and medical researchers to disclose protocols, anonymized subject-level data and study-level data when there is medical, scientific and/or public health interest to ensure the safe use of a Seqirus product licensed on or after 1 January 2014 in the United States (US) and/or the European Union (EU). This applies to Seqirus-sponsored interventional studies initiated after 27 September 2007 and ongoing as of 26 December 2007, that have been included as part of a US or EU submission package which received approval in US and EU on or after 1 January 2014 and have been accepted for publication
URL: https://www.seqirus.us/partnering

REFERENCES:
- [Background] Vesikari T, Karvonen A, Tilman S, Borkowski A, Montomoli E, Banzhoff A, Clemens R. Immunogenicity and safety of MF59-adjuvanted H5N1 influenza vaccine from infancy to adolescence. Pediatrics. 2010 Oct;126(4):e762-70. doi: 10.1542/peds.2009-2628. Epub 2010 Sep 6. PMID 20819892
- [Background] Vesikari T, Forsten A, Borkowski A, Gaitatzis N, Banzhoff A, Clemens R. Homologous and heterologous antibody responses to a one-year booster dose of an MF59((R)) adjuvanted A/H5N1 pre-pandemic influenza vaccine in pediatric subjects. Hum Vaccin Immunother. 2012 Jul;8(7):921-8. doi: 10.4161/hv.20248. Epub 2012 Jul 1. PMID 22777094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 2 centers in Estonia and 5 centers in the Philippines.
Pre-assignment Details: In total, 420 subjects were enrolled in the study.
Groups:
- Lowest Dose, Less Adjuvant aH5N1 Vaccine: 2 doses of lowest dose, less adjuvant aH5N1 by IM administration (Day 1 and Day 22)
- Low Dose, Less Adjuvant aH5N1 Vaccine: 2 doses of low dose, less adjuvant aH5N1 by IM administration (Day 1 and Day 22)
- Mid Dose, Less Adjuvant aH5N1 Vaccine: 2 doses of mid dose, less adjuvant aH5N1 by IM administration (Day 1 and Day 22)
- Lowest Dose, Adjuvanted aH5N1 Vaccine: 2 doses of lowest dose, adjuvanted aH5N1 by IM administration (Day 1 and Day 22)
- Low Dose, Adjuvanted aH5N1 Vaccine: 2 doses of low dose, adjuvanted aH5N1 by IM administration (Day 1 and Day 22)
- Mid Dose, Adjuvanted aH5N1 Vaccine: 2 doses of mid dose, adjuvanted aH5N1 by IM administration (Day 1 and Day 22)
Period: Overall Study
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Started | 69 | 72 | 70 | 70 | 69 | 70
Completed | 69 | 71 | 70 | 70 | 69 | 70
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine | Total
Number analyzed (Participants) | 69 | 72 | 70 | 70 | 69 | 70 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 69 | 72 | 70 | 70 | 69 | 70 | 420
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 48.2 (28.80) | 50.9 (31.61) | 47.1 (30.90) | 48.8 (31.81) | 49.9 (30.79) | 50.6 (31.77) | 49.3 (30.82)
Age, Customized [Count of Participants; unit: Participants]
  6 months to <36 months | 35 | 35 | 35 | 35 | 36 | 34 | 210
  3 years to <9 years | 34 | 37 | 35 | 35 | 33 | 36 | 210
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 33 | 31 | 31 | 40 | 192
  Male | 38 | 46 | 37 | 39 | 38 | 30 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 69 | 72 | 70 | 70 | 69 | 70 | 420
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 52 | 56 | 53 | 53 | 52 | 53 | 319
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 17 | 16 | 17 | 17 | 17 | 16 | 100
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Philippines | 52 | 56 | 53 | 53 | 52 | 54 | 320
  Estonia | 17 | 16 | 17 | 17 | 17 | 16 | 100
Received an influenza vaccination in the past 2 years [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 3 | 3 | 3 | 2 | 12
  No | 68 | 72 | 67 | 67 | 66 | 68 | 408

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint 1: Percentages of Subjects With Solicited Local and Systemic Adverse Events (AEs)
Description: Percentages of subjects with solicited local and systemic AEs that occurred within 7 days following each vaccination, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 through Day 7 and Day 22 through Day 28
Population: Solicited Safety Set, defined as all subjects in the All Exposed Set with any solicited AE data collected, including temperature measurements or use of analgesics/antipyretics.
  Results are presented for the overall study population and for the 6 months to <36 months and 3 years to <9 years age cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 69 | 72 | 70 | 70 | 69 | 70
Participants
  Solicited AEs (overall study population) | 32 | 33 | 32 | 34 | 37 | 31
  Solicited Local AEs (overall study population) | 19 | 16 | 16 | 21 | 19 | 17
  Solicited Systemic AEs (overall study population) | 21 | 24 | 20 | 24 | 29 | 18
  Analgesic/antipyretic use (overall study population) | 9 | 7 | 6 | 5 | 5 | 9
  Solicited AEs (6 months to <36 years age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Solicited AEs (6 months to <36 years age cohort) | 15 | 20 | 18 | 20 | 21 | 15
  Solicited Local AEs (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Solicited Local AEs (6 months to <36 months age cohort) | 7 | 10 | 6 | 11 | 8 | 4
  Solicited Systemic AEs (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Solicited Systemic AEs (6 months to <36 months age cohort) | 14 | 15 | 16 | 16 | 18 | 11
  Analgesic/antipyretic use (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Analgesic/antipyretic use (6 months to <36 months age cohort) | 5 | 4 | 4 | 3 | 3 | 6
  Solicited AEs (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Solicited AEs (3 years to <9 years age cohort) | 17 | 13 | 14 | 14 | 16 | 16
  Solicited Local AEs (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Solicited Local AEs (3 years to <9 years age cohort) | 12 | 6 | 10 | 10 | 11 | 13
  Solicited Systemic AEs (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Solicited Systemic AEs (3 years to <9 years age cohort) | 7 | 9 | 4 | 8 | 11 | 7
  Analgesic/antipyretic use (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Analgesic/antipyretic use (3 years to <9 years age cohort) | 4 | 3 | 2 | 2 | 2 | 3

2. Primary Outcome: Safety Endpoint 2: Percentages of Subjects With Any Unsolicited AEs
Description: Percentages of subjects with any unsolicited AEs reported within 21 days after each vaccination within each vaccine group, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 through Day 43
Population: Unsolicited Safety Set, defined as all subjects in the All Exposed Set with unsolicited AE data.
  Results are presented for the overall study population and for the 6 months to <36 months and 3 years to <9 years age cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 69 | 72 | 70 | 70 | 69 | 70
Participants
  Unsolicited AEs, Any (overall study population) | 18 | 15 | 20 | 10 | 15 | 12
  Unsolicited AEs, Mild (overall study population) | 18 | 14 | 20 | 10 | 12 | 9
  Unsolicited AEs, Moderate (overall study population) | 0 | 1 | 0 | 0 | 3 | 2
  Unsolicited AEs, Severe (overall study population) | 0 | 0 | 0 | 0 | 0 | 1
  Unsolicited AEs, Related (overall study population) | 2 | 2 | 2 | 0 | 2 | 1
  Unsolicited AEs, Any (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Unsolicited AEs, Any (6 months to <36 months age cohort) | 12 | 11 | 13 | 8 | 8 | 7
  Unsolicited AEs, Mild (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Unsolicited AEs, Mild (6 months to <36 months age cohort) | 12 | 10 | 13 | 8 | 7 | 5
  Unsolicited AEs, Moderate (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Unsolicited AEs, Moderate (6 months to <36 months age cohort) | 0 | 1 | 0 | 0 | 1 | 2
  Unsolicited AEs, Severe (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Unsolicited AEs, Severe (6 months to <36 months age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  Unsolicited AEs, Related (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Unsolicited AEs, Related (6 months to <36 months age cohort) | 1 | 2 | 2 | 0 | 1 | 0
  Unsolicited AEs, Any (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Unsolicited AEs, Any (3 years to <9 years age cohort) | 6 | 4 | 7 | 2 | 7 | 5
  Unsolicited AEs, Mild (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Unsolicited AEs, Mild (3 years to <9 years age cohort) | 6 | 4 | 7 | 2 | 5 | 4
  Unsolicited AEs, Moderate (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Unsolicited AEs, Moderate (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 2 | 0
  Unsolicited AEs, Severe (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Unsolicited AEs, Severe (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 0 | 1
  Unsolicited AEs, Related (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Unsolicited AEs, Related (3 years to <9 years age cohort) | 1 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Safety Endpoint 3: Percentages of Subjects Reporting Serious Adverse Events (SAEs), New-onset Chronic Disease (NOCD), Adverse Events of Special Interest (AESI), and AEs Leading to Vaccine and/or Study Withdrawal
Description: Percentages of subjects reporting SAEs, NOCDs, AESIs, and AEs leading to vaccine and/or study withdrawal, as collected from Day 1 through Day 387, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 through Day 387
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 69 | 72 | 70 | 70 | 69 | 70
Participants
  SAE (overall study population) | 0 | 1 | 3 | 0 | 1 | 3
  Related SAE (overall study population) | 0 | 0 | 0 | 0 | 0 | 0
  NOCD (overall study population) | 0 | 1 | 0 | 0 | 0 | 0
  AESI (overall study population) | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to withdrawal (overall study population) | 0 | 0 | 0 | 0 | 0 | 0
  Death (overall study population) | 0 | 1 | 0 | 0 | 0 | 0
  SAE (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  SAE (6 months to <36 months age cohort) | 0 | 1 | 1 | 0 | 1 | 2
  Related SAE (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Related SAE (6 months to <36 months age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  NOCD (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  NOCD (6 months to <36 months age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  AESI (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  AESI (6 months to <36 months age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to withdrawal (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  AE leading to withdrawal (6 months to <36 months age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  Death (6 months to <36 months age cohort): number analyzed (Participants) | 35 | 35 | 35 | 35 | 36 | 34
  Death (6 months to <36 months age cohort) | 0 | 1 | 0 | 0 | 0 | 0
  SAE (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  SAE (3 years to <9 years age cohort) | 0 | 0 | 2 | 0 | 0 | 1
  Related SAE (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Related SAE (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  NOCD (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  NOCD (3 years to <9 years age cohort) | 0 | 1 | 0 | 0 | 0 | 0
  AESI (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  AESI (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  AE leading to withdrawal (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  AE leading to withdrawal (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 0 | 0
  Death (3 years to <9 years age cohort): number analyzed (Participants) | 34 | 37 | 35 | 35 | 33 | 36
  Death (3 years to <9 years age cohort) | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Primary Immunogenicity Endpoint 1a: Geometric Mean Titers (GMTs), as Measured by Hemagglutination Inhibition (HI) and Microneutralization (MN) Assays Against the Homologous H5N1 Strain
Description: GMTs on Day 1 (prior to the first vaccination), Day 22 (3 weeks after the first vaccination), and Day 43 (3 weeks after the second vaccination) as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 (baseline), Day 22, and Day 43
Population: Per Protocol Set (PPS) Immunogenicity, defined as all subjects in the Full Analysis Set (FAS) Immunogenicity who: correctly received the vaccine; provided at least the baseline and one postbaseline blood sample, with evaluable immunogenicity data; had no protocol deviations leading to exclusion as defined prior to unblinding/analysis.
  Results are presented for the overall study population and for the 6 months to <36 months and 3 years to <9 years age cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
titer
  HI GMT Day 1 (overall study population) | 5.05 [4.8 to 5.3] | 5.00 [4.8 to 5.2] | 5.21 [5.0 to 5.4] | 5.05 [4.8 to 5.3] | 5.00 [4.8 to 5.2] | 5.24 [5.0 to 5.5]
  HI GMT Day 22 (overall study population) | 5.61 [4.9 to 6.4] | 6.21 [5.5 to 7.0] | 5.98 [5.3 to 6.8] | 6.17 [5.4 to 7.0] | 6.47 [5.7 to 7.3] | 5.78 [5.1 to 6.6]
  HI GMT Day 43 (overall study population) | 81.10 [58.3 to 112.8] | 68.06 [49.4 to 93.8] | 86.70 [62.3 to 120.7] | 122.43 [87.8 to 170.7] | 123.37 [89.1 to 170.8] | 123.61 [88.8 to 172.1]
  HI GMT Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMT Day 1 (6 months to <36 months age cohort) | 5.10 [4.9 to 5.3] | 5.00 [4.8 to 5.2] | 5.42 [5.2 to 5.7] | 5.11 [4.9 to 5.3] | 5.00 [4.8 to 5.2] | 5.00 [4.8 to 5.2]
  HI GMT Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMT Day 22 (6 months to <36 months age cohort) | 5.59 [4.7 to 6.6] | 6.14 [5.2 to 7.3] | 5.51 [4.6 to 6.6] | 6.23 [5.2 to 7.4] | 6.55 [5.5 to 7.8] | 5.78 [4.8 to 6.9]
  HI GMT Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMT Day 43 (6 months to <36 months age cohort) | 93.22 [56.5 to 153.7] | 98.37 [59.6 to 162.4] | 102.28 [61.5 to 170.1] | 129.72 [78.1 to 215.5] | 157.44 [96.7 to 256.3] | 120.07 [71.0 to 202.9]
  HI GMT Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMT Day 1 (3 years to <9 years age cohort) | 5.00 [4.6 to 5.4] | 5.00 [4.7 to 5.4] | 5.00 [4.6 to 5.4] | 5.00 [4.6 to 5.4] | 5.00 [4.6 to 5.4] | 5.45 [5.1 to 5.9]
  HI GMT Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMT Day 22 (3 years to <9 years age cohort) | 5.61 [4.6 to 6.8] | 6.32 [5.3 to 7.6] | 6.29 [5.2 to 7.6] | 6.10 [5.0 to 7.4] | 6.42 [5.3 to 7.8] | 5.91 [4.9 to 7.1]
  HI GMT Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMT Day 43 (3 years to <9 years age cohort) | 70.21 [45.5 to 108.4] | 48.35 [32.1 to 72.9] | 69.40 [44.9 to 107.2] | 114.85 [74.4 to 177.4] | 97.17 [62.9 to 150.1] | 129.15 [84.9 to 196.6]
  MN GMT Day 1 (overall study population) | 5.19 [4.9 to 5.5] | 5.27 [5.0 to 5.6] | 5.38 [5.1 to 5.7] | 5.16 [4.9 to 5.5] | 5.13 [4.9 to 5.4] | 5.31 [5.0 to 5.6]
  MN GMT Day 22 (overall study population): number analyzed (Participants) | 67 | 69 | 67 | 64 | 66 | 67
  MN GMT Day 22 (overall study population) | 31.42 [24.7 to 40.0] | 34.83 [27.5 to 44.2] | 40.61 [31.9 to 51.7] | 46.08 [36.0 to 59.0] | 54.66 [42.9 to 69.7] | 52.81 [41.5 to 67.2]
  MN GMT Day 43 (overall study population): number analyzed (Participants) | 67 | 70 | 67 | 66 | 69 | 67
  MN GMT Day 43 (overall study population) | 531.04 [424.7 to 664.1] | 667.86 [536.7 to 831.1] | 610.37 [488.0 to 763.4] | 619.44 [494.5 to 775.9] | 864.91 [693.8 to 1078.2] | 766.18 [612.6 to 958.2]
  MN GMT Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMT Day 1 (6 months to <36 months age cohort) | 5.00 [4.7 to 5.3] | 5.00 [4.7 to 5.3] | 5.26 [4.9 to 5.6] | 5.21 [4.9 to 5.6] | 5.10 [4.8 to 5.4] | 5.29 [4.9 to 5.7]
  MN GMT Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 31 | 34 | 31
  MN GMT Day 22 (6 months to <36 months age cohort) | 29.27 [21.0 to 40.8] | 33.14 [23.8 to 46.2] | 24.93 [17.9 to 34.7] | 45.78 [32.3 to 64.8] | 69.41 [49.8 to 96.7] | 42.07 [29.7 to 59.6]
  MN GMT Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMT Day 43 (6 months to <36 months age cohort) | 618.77 [448.2 to 854.3] | 910.32 [659.3 to 1256.9] | 717.83 [520.0 to 991.0] | 725.06 [522.8 to 1005.5] | 1094.07 [800.0 to 1496.2] | 863.94 [616.3 to 1211.2]
  MN GMT Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  MN GMT Day 1 (3 years to <9 years age cohort) | 5.38 [4.9 to 5.9] | 5.54 [5.1 to 6.0] | 5.49 [5.0 to 6.0] | 5.11 [4.7 to 5.6] | 5.16 [4.7 to 5.7] | 5.35 [4.9 to 5.8]
  MN GMT Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 35 | 33 | 33 | 32 | 36
  MN GMT Day 22 (3 years to <9 years age cohort) | 33.70 [24.0 to 47.4] | 36.69 [26.3 to 51.1] | 66.97 [47.6 to 94.2] | 46.59 [33.1 to 65.6] | 42.11 [29.8 to 59.6] | 65.11 [47.0 to 90.2]
  MN GMT Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 36 | 33 | 33 | 33 | 36
  MN GMT Day 43 (3 years to <9 years age cohort) | 458.11 [334.2 to 627.9] | 495.77 [366.4 to 670.9] | 518.46 [378.2 to 710.8] | 527.09 [384.3 to 723.0] | 680.71 [496.4 to 933.4] | 670.67 [495.9 to 907.0]

5. Primary Outcome: Primary Immunogenicity Endpoint 1b: Geometric Mean Ratios (GMR), as Measured by HI and MN Assays Against the Homologous H5N1 Strain
Description: GMRs calculated as follows: Day 22/Day 1 and Day 43/Day 1 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 (baseline), Day 22, and Day 43
Population: PPS Immunogenicity, defined as all subjects in the FAS Immunogenicity who: correctly received the vaccine; provided at least the baseline and one postbaseline blood sample, with evaluable immunogenicity data; had no protocol deviations leading to exclusion as defined prior to unblinding/analysis.
  Results are presented for the overall study population and for the 6 months to <36 months and 3 years to <9 years age cohorts.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
ratio
  HI GMR Day 22/Day 1 (overall study population) | 1.11 [1.0 to 1.3] | 1.24 [1.1 to 1.4] | 1.15 [1.0 to 1.3] | 1.22 [1.1 to 1.4] | 1.29 [1.1 to 1.5] | 1.11 [1.0 to 1.3]
  HI GMR Day 43/Day 1 (overall study population) | 16.14 [11.5 to 22.6] | 13.77 [9.9 to 19.1] | 16.38 [11.7 to 23.0] | 24.35 [17.3 to 34.2] | 24.98 [17.9 to 34.8] | 23.14 [16.5 to 32.4]
  HI GMR Day 22/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMR Day 22/Day 1 (6 months to <36 months age cohort) | 1.10 [0.9 to 1.3] | 1.21 [1.0 to 1.4] | 1.05 [0.9 to 1.3] | 1.22 [1.0 to 1.5] | 1.30 [1.1 to 1.5] | 1.14 [1.0 to 1.4]
  HI GMR Day 43/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMR Day 43/Day 1 (6 months to <36 months age cohort) | 18.27 [11.1 to 30.1] | 19.62 [11.9 to 32.4] | 19.02 [11.5 to 31.4] | 25.41 [15.3 to 42.2] | 31.39 [19.3 to 51.1] | 23.94 [14.2 to 40.4]
  HI GMR Day 22/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMR Day 22/Day 1 (3 years to <9 years age cohort) | 1.12 [0.9 to 1.4] | 1.26 [1.0 to 1.5] | 1.26 [1.0 to 1.5] | 1.22 [1.0 to 1.5] | 1.29 [1.0 to 1.6] | 1.08 [0.9 to 1.3]
  HI GMR Day 43/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMR Day 43/Day 1 (3 years to <9 years age cohort) | 14.27 [9.0 to 22.6] | 9.83 [6.4 to 15.2] | 14.10 [8.9 to 22.3] | 23.34 [14.7 to 37.0] | 19.75 [12.5 to 31.3] | 21.98 [14.2 to 34.1]
  MN GMR Day 22/Day 1 (overall study population): number analyzed (Participants) | 67 | 69 | 67 | 64 | 66 | 67
  MN GMR Day 22/Day 1 (overall study population) | 6.02 [4.7 to 7.7] | 6.62 [5.2 to 8.4] | 7.66 [6.0 to 9.8] | 8.85 [6.9 to 11.3] | 10.52 [8.2 to 13.4] | 10.02 [7.9 to 12.8]
  MN GMR Day 43/Day 1 (overall study population): number analyzed (Participants) | 67 | 70 | 67 | 66 | 69 | 67
  MN GMR Day 43/Day 1 (overall study population) | 102.26 [81.4 to 128.5] | 126.71 [101.4 to 158.4] | 113.98 [90.7 to 143.2] | 119.78 [95.2 to 150.7] | 168.06 [134.2 to 210.5] | 144.55 [115.0 to 181.6]
  MN GMR Day 22/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 31 | 34 | 31
  MN GMR Day 22/Day 1 (6 months to <36 months age cohort) | 5.76 [4.1 to 8.0] | 6.52 [4.7 to 9.1] | 4.80 [3.4 to 6.7] | 8.84 [6.2 to 12.5] | 13.54 [9.7 to 18.9] | 8.09 [5.7 to 11.4]
  MN GMR Day 43/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMR Day 43/Day 1 (6 months to <36 months age cohort) | 122.81 [88.8 to 169.9] | 180.68 [130.6 to 250.0] | 137.36 [99.3 to 190.0] | 139.62 [100.4 to 194.1] | 214.16 [156.2 to 293.6] | 164.74 [117.3 to 231.4]
  MN GMR Day 22/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 35 | 33 | 33 | 32 | 36
  MN GMR Day 22/Day 1 (3 years to <9 years age cohort) | 6.29 [4.5 to 8.9] | 6.73 [4.8 to 9.4] | 12.37 [8.8 to 17.4] | 8.90 [6.3 to 12.5] | 8.00 [5.7 to 11.3] | 12.18 [8.8 to 16.9]
  MN GMR Day 43/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 36 | 33 | 33 | 33 | 36
  MN GMR Day 43/Day 1 (3 years to <9 years age cohort) | 85.22 [61.6 to 118.0] | 89.57 [65.6 to 122.3] | 94.64 [68.4 to 131.0] | 102.76 [74.2 to 142.3] | 131.50 [95.0 to 182.0] | 125.44 [91.9 to 171.3]

6. Primary Outcome: Primary Immunogenicity Endpoint 1c: Percentage of Subjects Achieving Seroconversion (Non-detectable to ≥1:40, or 4-fold Increase From a Detectable Day 1 Titer)
Description: Percentage of subjects achieving seroconversion (non-detectable to ≥1:40, or 4-fold increase from a detectable Day 1 titer) on Day 22 and Day 43 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 (baseline), Day 22, and Day 43
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
percentage of participants
  HI seroconversion at Day 22 (overall study population) | 0.0 [0.00 to 5.36] | 4.2 [0.88 to 11.86] | 3.0 [0.36 to 10.37] | 4.5 [0.95 to 12.71] | 1.4 [0.04 to 7.81] | 3.0 [0.36 to 10.37]
  HI seroconversion at Day 43 (overall study population) | 82.1 [70.80 to 90.39] | 74.6 [62.92 to 84.23] | 77.6 [65.78 to 86.89] | 90.9 [81.26 to 96.59] | 87.0 [76.68 to 93.86] | 86.6 [76.03 to 93.67]
  HI seroconversion at Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI seroconversion at Day 22 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 2.9 [0.07 to 15.33] | 0.0 [0.00 to 10.28] | 3.0 [0.08 to 15.76] | 0.0 [0.00 to 9.74] | 3.2 [0.08 to 16.70]
  HI seroconversion at Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI seroconversion at Day 43 (6 months to <36 months age cohort) | 79.4 [62.10 to 91.30] | 82.4 [65.47 to 93.24] | 79.4 [62.10 to 91.30] | 93.9 [79.77 to 99.26] | 86.1 [70.50 to 95.33] | 87.1 [70.17 to 96.37]
  HI seroconversion at Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI seroconversion at Day 22 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 5.4 [0.66 to 18.19] | 6.1 [0.74 to 20.23] | 6.1 [0.74 to 20.23] | 3.0 [0.08 to 15.76] | 2.8 [0.07 to 14.53]
  HI seroconversion at Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI seroconversion at Day 43 (3 years to <9 years age cohort) | 84.8 [68.10 to 94.89] | 67.6 [50.21 to 81.99] | 75.8 [57.74 to 88.91] | 87.9 [71.80 to 96.60] | 87.9 [71.80 to 96.60] | 86.1 [70.50 to 95.33]
  MN seroconversion at Day 22 (overall study population): number analyzed (Participants) | 67 | 69 | 67 | 64 | 66 | 67
  MN seroconversion at Day 22 (overall study population) | 44.8 [32.60 to 57.42] | 56.5 [44.04 to 68.42] | 58.2 [45.52 to 70.15] | 67.2 [54.31 to 78.41] | 72.7 [60.36 to 82.97] | 68.7 [56.16 to 79.44]
  MN seroconversion at Day 43 (overall study population): number analyzed (Participants) | 67 | 70 | 67 | 66 | 69 | 67
  MN seroconversion at Day 43 (overall study population) | 100.0 [94.64 to 100.00] | 100.0 [94.87 to 100.00] | 100.0 [94.64 to 100.00] | 100.0 [94.56 to 100.00] | 100.0 [94.79 to 100.00] | 100.0 [94.64 to 100.00]
  MN seroconversion at Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 31 | 34 | 31
  MN seroconversion at Day 22 (6 months to <36 months age cohort) | 35.3 [19.75 to 53.51] | 55.9 [37.89 to 72.81] | 35.3 [19.75 to 53.51] | 71.0 [51.96 to 85.78] | 82.4 [65.47 to 93.24] | 58.1 [39.08 to 75.45]
  MN seroconversion at Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN seroconversion at Day 43 (6 months to <36 months age cohort) | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00] | 100.0 [88.78 to 100.00]
  MN seroconversion at Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 35 | 33 | 33 | 32 | 36
  MN seroconversion at Day 22 (3 years to <9 years age cohort) | 54.5 [36.35 to 71.89] | 57.1 [39.35 to 73.68] | 81.8 [64.54 to 93.02] | 63.6 [45.12 to 79.60] | 62.5 [43.69 to 78.90] | 77.8 [60.85 to 89.88]
  MN seroconversion at Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 36 | 33 | 33 | 33 | 36
  MN seroconversion at Day 43 (3 years to <9 years age cohort) | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00]

7. Primary Outcome: Primary Immunogenicity Endpoint 1d: Percentage of Subjects Achieving Seroconversion With a Titer ≥1:40
Description: Percentage of subjects achieving seroconversion with a titer ≥1:40 on Day 1, Day 22, and Day 43 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
  No statistical analyses have been specified for this primary endpoint. The statistical analysis was descriptive in nature without any prespecified inferential analyses.
Time Frame: Day 1 (baseline), Day 22, and Day 43
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
percentage of participants
  HI titer ≥1:40 at Day 1 (overall study population) | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.06] | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.44] | 0.0 [0.00 to 5.21] | 1.5 [0.04 to 8.04]
  HI titer ≥1:40 at Day 22 (overall study population) | 0.0 [0.00 to 5.36] | 4.2 [0.88 to 11.86] | 3.0 [0.36 to 10.37] | 4.5 [0.95 to 12.71] | 1.4 [0.04 to 7.81] | 3.0 [0.36 to 10.37]
  HI titer ≥1:40 at Day 43 (overall study population) | 82.1 [70.80 to 90.39] | 74.6 [62.92 to 84.23] | 77.6 [65.78 to 86.89] | 90.9 [81.26 to 96.59] | 87.0 [76.68 to 93.86] | 86.6 [76.03 to 93.67]
  HI titer ≥1:40 at Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI titer ≥1:40 at Day 1 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74] | 0.0 [0.00 to 11.22]
  HI titer ≥1:40 at Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI titer ≥1:40 at Day 22 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 2.9 [0.07 to 15.33] | 0.0 [0.00 to 10.28] | 3.0 [0.08 to 15.76] | 0.0 [0.00 to 9.74] | 3.2 [0.08 to 16.70]
  HI titer ≥1:40 at Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI titer ≥1:40 at Day 43 (6 months to <36 months age cohort) | 79.4 [62.10 to 91.30] | 82.4 [65.47 to 93.24] | 79.4 [62.10 to 91.30] | 93.9 [79.77 to 99.26] | 86.1 [70.50 to 95.33] | 87.1 [70.17 to 96.37]
  HI titer ≥1:40 at Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI titer ≥1:40 at Day 1 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.49] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 2.8 [0.07 to 14.53]
  HI titer ≥1:40 at Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI titer ≥1:40 at Day 22 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 5.4 [0.66 to 18.19] | 6.1 [0.74 to 20.23] | 6.1 [0.74 to 20.23] | 3.0 [0.08 to 15.76] | 2.8 [0.07 to 14.53]
  HI titer ≥1:40 at Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI titer ≥1:40 at Day 43 (3 years to <9 years age cohort) | 84.8 [68.10 to 94.89] | 67.6 [50.21 to 81.99] | 75.8 [57.74 to 88.91] | 87.9 [71.80 to 96.60] | 87.9 [71.80 to 96.60] | 86.1 [70.50 to 95.33]
  MN titer ≥1:40 at Day 1 (overall study population) | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.06] | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.44] | 0.0 [0.00 to 5.21] | 0.0 [0.00 to 5.36]
  MN titer ≥1:40 at Day 22 (overall study population): number analyzed (Participants) | 67 | 69 | 67 | 64 | 66 | 67
  MN titer ≥1:40 at Day 22 (overall study population) | 44.8 [32.60 to 57.42] | 56.5 [44.04 to 68.42] | 58.2 [45.52 to 70.15] | 67.2 [54.31 to 78.41] | 72.7 [60.36 to 82.97] | 68.7 [56.16 to 79.44]
  MN titer ≥1:40 at Day 43 (overall study population): number analyzed (Participants) | 67 | 70 | 67 | 66 | 69 | 67
  MN titer ≥1:40 at Day 43 (overall study population) | 100.0 [94.64 to 100.00] | 100.0 [94.87 to 100.00] | 100.0 [94.64 to 100.00] | 100.0 [94.56 to 100.00] | 100.0 [94.79 to 100.00] | 100.0 [94.64 to 100.00]
  MN titer ≥1:40 at Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN titer ≥1:40 at Day 1 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74] | 0.0 [0.00 to 11.22]
  MN titer ≥1:40 at Day 22 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 31 | 34 | 31
  MN titer ≥1:40 at Day 22 (6 months to <36 months age cohort) | 35.3 [19.75 to 53.51] | 55.9 [37.89 to 72.81] | 35.3 [19.75 to 53.51] | 71.0 [51.96 to 85.78] | 82.4 [65.47 to 93.24] | 58.1 [39.08 to 75.45]
  MN titer ≥1:40 at Day 43 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN titer ≥1:40 at Day 43 (6 months to <36 months age cohort) | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00] | 100.0 [88.78 to 100.00]
  MN titer ≥1:40 at Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  MN titer ≥1:40 at Day 1 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.49] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74]
  MN titer ≥1:40 at Day 22 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 35 | 33 | 33 | 32 | 36
  MN titer ≥1:40 at Day 22 (3 years to <9 years age cohort) | 54.5 [36.35 to 71.89] | 57.1 [39.35 to 73.68] | 81.8 [64.54 to 93.02] | 63.6 [45.12 to 79.60] | 62.5 [43.69 to 78.90] | 77.8 [60.85 to 89.88]
  MN titer ≥1:40 at Day 43 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 36 | 33 | 33 | 33 | 36
  MN titer ≥1:40 at Day 43 (3 years to <9 years age cohort) | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [89.42 to 100.00] | 100.0 [90.26 to 100.00]

8. Secondary Outcome: Secondary Immunogenicity Endpoint 1a: GMTs, as Measured by HI and MN Assays Against the Homologous H5N1 Strain
Description: GMTs on Day 1 (prior to the first vaccination) and Day 202 (6 months after the second vaccination) as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
Time Frame: Day 1 (baseline) and Day 202
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
titer
  HI GMT Day 1 (overall study population) | 5.05 [4.8 to 5.3] | 5.00 [4.8 to 5.2] | 5.21 [5.0 to 5.4] | 5.05 [4.8 to 5.3] | 5.00 [4.8 to 5.2] | 5.24 [5.0 to 5.5]
  HI GMT Day 202 (overall study population) | 7.92 [6.3 to 9.9] | 8.90 [7.2 to 11.0] | 8.81 [7.1 to 11.0] | 10.19 [8.2 to 12.7] | 12.90 [10.4 to 16.1] | 13.15 [10.5 to 16.4]
  HI GMT Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMT Day 1 (6 months to <36 months age cohort) | 5.10 [4.9 to 5.3] | 5.00 [4.8 to 5.2] | 5.42 [5.2 to 5.7] | 5.11 [4.9 to 5.3] | 5.00 [4.8 to 5.2] | 5.00 [4.8 to 5.2]
  HI GMT Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMT Day 202 (6 months to <36 months age cohort) | 9.11 [6.3 to 13.3] | 12.57 [8.6 to 18.3] | 11.60 [7.9 to 17.0] | 13.55 [9.3 to 19.8] | 19.12 [13.3 to 27.6] | 19.00 [12.8 to 28.2]
  HI GMT Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMT Day 1 (3 years to <9 years age cohort) | 5.00 [4.6 to 5.4] | 5.00 [4.7 to 5.4] | 5.00 [4.6 to 5.4] | 5.00 [4.6 to 5.4] | 5.00 [4.6 to 5.4] | 5.45 [5.1 to 5.9]
  HI GMT Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMT Day 202 (3 years to <9 years age cohort) | 6.90 [5.4 to 8.8] | 6.36 [5.1 to 8.0] | 6.55 [5.2 to 8.3] | 7.66 [6.0 to 9.7] | 8.69 [6.8 to 11.0] | 9.30 [7.4 to 11.7]
  MN GMT Day 1 (overall study population) | 5.19 [4.9 to 5.5] | 5.27 [5.0 to 5.6] | 5.38 [5.1 to 5.7] | 5.16 [4.9 to 5.5] | 5.13 [4.9 to 5.4] | 5.31 [5.0 to 5.6]
  MN GMT Day 202 (overall study population): number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 66
  MN GMT Day 202 (overall study population) | 113.24 [94.7 to 135.4] | 146.98 [123.6 to 174.8] | 146.41 [122.4 to 175.1] | 150.56 [125.7 to 180.3] | 183.15 [153.6 to 218.4] | 195.57 [163.3 to 234.2]
  MN GMT Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMT Day 1 (6 months to <36 months age cohort) | 5.00 [4.7 to 5.3] | 5.00 [4.7 to 5.3] | 5.26 [4.9 to 5.6] | 5.21 [4.9 to 5.6] | 5.10 [4.8 to 5.4] | 5.29 [4.9 to 5.7]
  MN GMT Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMT Day 202 (6 months to <36 months age cohort) | 144.60 [111.8 to 187.0] | 217.84 [168.4 to 281.7] | 175.31 [135.6 to 226.7] | 174.21 [134.2 to 226.1] | 245.52 [191.3 to 315.1] | 268.31 [205.0 to 351.3]
  MN GMT Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  MN GMT Day 1 (3 years to <9 years age cohort) | 5.38 [4.9 to 5.9] | 5.54 [5.1 to 6.0] | 5.49 [5.0 to 6.0] | 5.11 [4.7 to 5.6] | 5.16 [4.7 to 5.7] | 5.35 [4.9 to 5.8]
  MN GMT Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 35
  MN GMT Day 202 (3 years to <9 years age cohort) | 89.38 [69.6 to 114.8] | 101.19 [79.8 to 128.2] | 122.19 [95.1 to 157.0] | 129.11 [100.4 to 165.9] | 136.08 [105.9 to 174.9] | 142.59 [111.8 to 181.8]

9. Secondary Outcome: Secondary Immunogenicity Endpoint 1b: GMRs, as Measured by HI and MN Assays Against the Homologous H5N1 Strain
Description: GMRs calculated as follows: Day 202/Day 1 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
Time Frame: Day 1 (baseline) and Day 202
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
ratio
  HI GMR Day 202/Day 1 (overall study population) | 1.57 [1.3 to 2.0] | 1.78 [1.4 to 2.2] | 1.69 [1.3 to 2.1] | 2.02 [1.6 to 2.5] | 2.59 [2.1 to 3.2] | 2.50 [2.0 to 3.1]
  HI GMR Day 202/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI GMR Day 202/Day 1 (6 months to <36 months age cohort) | 1.79 [1.2 to 2.6] | 2.50 [1.7 to 3.6] | 2.17 [1.5 to 3.2] | 2.65 [1.8 to 3.9] | 3.81 [2.6 to 5.5] | 3.78 [2.5 to 5.6]
  HI GMR Day 202/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI GMR Day 202/Day 1 (3 years to <9 years age cohort) | 1.38 [1.1 to 1.8] | 1.28 [1.0 to 1.6] | 1.31 [1.0 to 1.7] | 1.54 [1.2 to 2.0] | 1.74 [1.4 to 2.2] | 1.68 [1.3 to 2.1]
  MN GMR Day 202/Day 1 (overall study population): number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 66
  MN GMR Day 202/Day 1 (overall study population) | 21.77 [18.1 to 26.1] | 27.94 [23.4 to 33.4] | 27.45 [22.9 to 33.0] | 29.04 [24.2 to 34.9] | 35.47 [29.6 to 42.5] | 36.95 [30.7 to 44.4]
  MN GMR Day 202/Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN GMR Day 202/Day 1 (6 months to <36 months age cohort) | 28.49 [22.0 to 36.9] | 42.91 [33.2 to 55.5] | 33.76 [26.1 to 43.7] | 33.68 [25.9 to 43.7] | 47.95 [37.3 to 61.6] | 51.56 [39.4 to 67.5]
  MN GMR Day 202/Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 35
  MN GMR Day 202/Day 1 (3 years to <9 years age cohort) | 16.64 [12.8 to 21.6] | 18.41 [14.4 to 23.5] | 22.38 [17.3 to 29.0] | 25.04 [19.3 to 32.5] | 26.18 [20.2 to 34.0] | 26.63 [20.7 to 34.3]

10. Secondary Outcome: Secondary Immunogenicity Endpoint 1c: Percentage of Subjects Achieving Seroconversion (Non-detectable to ≥1:40, or 4-fold Increase From a Detectable Day 1 Titer)
Description: Percentage of subjects achieving seroconversion (non-detectable to ≥1:40, or 4-fold increase from a detectable Day 1 titer) on Day 202 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
Time Frame: Day 1 (baseline) and Day 202
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
percentage of participants
  HI seroconversion at Day 202 (overall study population) | 10.4 [4.30 to 20.35] | 14.1 [6.97 to 24.38] | 11.9 [5.30 to 22.18] | 15.2 [7.51 to 26.10] | 21.7 [12.71 to 33.31] | 25.4 [15.53 to 37.49]
  HI seroconversion at Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI seroconversion at Day 202 (6 months to <36 months age cohort) | 17.6 [6.76 to 34.53] | 26.5 [12.88 to 44.36] | 23.5 [10.75 to 41.17] | 27.3 [13.30 to 45.52] | 33.3 [18.56 to 50.97] | 41.9 [24.55 to 60.92]
  HI seroconversion at Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI seroconversion at Day 202 (3 years to <9 years age cohort) | 3.0 [0.08 to 15.76] | 2.7 [0.07 to 14.16] | 0.0 [0.00 to 10.58] | 3.0 [0.08 to 15.76] | 9.1 [1.92 to 24.33] | 11.1 [3.11 to 26.06]
  MN seroconversion at Day 202 (overall study population): number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 66
  MN seroconversion at Day 202 (overall study population) | 95.5 [87.47 to 99.07] | 97.2 [90.19 to 99.66] | 100.0 [94.64 to 100.00] | 97.0 [89.48 to 99.63] | 98.6 [92.19 to 99.96] | 97.0 [89.48 to 99.63]
  MN seroconversion at Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN seroconversion at Day 202 (6 months to <36 months age cohort) | 97.1 [84.67 to 99.93] | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 97.0 [84.24 to 99.92] | 100.0 [90.26 to 100.00] | 100.0 [88.78 to 100.00]
  MN seroconversion at Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 35
  MN seroconversion at Day 202 (3 years to <9 years age cohort) | 93.9 [79.77 to 99.26] | 94.6 [81.81 to 99.34] | 100.0 [89.42 to 100.00] | 97.0 [84.24 to 99.92] | 97.0 [84.24 to 99.92] | 94.3 [80.84 to 99.30]

11. Secondary Outcome: Secondary Immunogenicity Endpoint 1d: Percentage of Subjects Achieving Seroconversion With a Titer ≥1:40
Description: Percentage of subjects achieving seroconversion with a titer ≥1:40 on Day 1 and Day 202 as determined by HI and MN assays against the homologous H5N1 pandemic influenza strain, by total population and by age cohort.
Time Frame: Day 1 (baseline) and Day 202
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
Number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 67
percentage of participants
  HI titer ≥1:40 at Day 1 (overall study population) | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.06] | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.44] | 0.0 [0.00 to 5.21] | 1.5 [0.04 to 8.04]
  HI titer ≥1:40 at Day 202 (overall study population) | 10.4 [4.30 to 20.35] | 14.1 [6.97 to 24.38] | 11.9 [5.30 to 22.18] | 15.2 [7.51 to 26.10] | 21.7 [12.71 to 33.31] | 25.4 [15.53 to 37.49]
  HI titer ≥1:40 at Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI titer ≥1:40 at Day 1 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74] | 0.0 [0.00 to 11.22]
  HI titer ≥1:40 at Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  HI titer ≥1:40 at Day 202 (6 months to <36 months age cohort) | 17.6 [6.76 to 34.53] | 26.5 [12.88 to 44.36] | 23.5 [10.75 to 41.17] | 27.3 [13.30 to 45.52] | 33.3 [18.56 to 50.97] | 41.9 [24.55 to 60.92]
  HI titer ≥1:40 at Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI titer ≥1:40 at Day 1 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.49] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 2.8 [0.07 to 14.53]
  HI titer ≥1:40 at Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  HI titer ≥1:40 at Day 202 (3 years to <9 years age cohort) | 3.0 [0.08 to 15.76] | 2.7 [0.07 to 14.16] | 0.0 [0.00 to 10.58] | 3.0 [0.08 to 15.76] | 9.1 [1.92 to 24.33] | 11.1 [3.11 to 26.06]
  MN titer ≥1:40 at Day 1 (overall study population) | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.06] | 0.0 [0.00 to 5.36] | 0.0 [0.00 to 5.44] | 0.0 [0.00 to 5.21] | 0.0 [0.00 to 5.36]
  MN titer ≥1:40 at Day 202 (overall study population): number analyzed (Participants) | 67 | 71 | 67 | 66 | 69 | 66
  MN titer ≥1:40 at Day 202 (overall study population) | 95.5 [87.47 to 99.07] | 98.6 [92.40 to 99.96] | 100.0 [94.64 to 100.00] | 97.0 [89.48 to 99.63] | 98.6 [92.19 to 99.96] | 98.5 [91.84 to 99.96]
  MN titer ≥1:40 at Day 1 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN titer ≥1:40 at Day 1 (6 months to <36 months age cohort) | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.28] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74] | 0.0 [0.00 to 11.22]
  MN titer ≥1:40 at Day 202 (6 months to <36 months age cohort): number analyzed (Participants) | 34 | 34 | 34 | 33 | 36 | 31
  MN titer ≥1:40 at Day 202 (6 months to <36 months age cohort) | 97.1 [84.67 to 99.93] | 100.0 [89.72 to 100.00] | 100.0 [89.72 to 100.00] | 97.0 [84.24 to 99.92] | 100.0 [90.26 to 100.00] | 100.0 [88.78 to 100.00]
  MN titer ≥1:40 at Day 1 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 36
  MN titer ≥1:40 at Day 1 (3 years to <9 years age cohort) | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.49] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 10.58] | 0.0 [0.00 to 9.74]
  MN titer ≥1:40 at Day 202 (3 years to <9 years age cohort): number analyzed (Participants) | 33 | 37 | 33 | 33 | 33 | 35
  MN titer ≥1:40 at Day 202 (3 years to <9 years age cohort) | 93.9 [79.77 to 99.26] | 97.3 [85.84 to 99.93] | 100.0 [89.42 to 100.00] | 97.0 [84.24 to 99.92] | 97.0 [84.24 to 99.92] | 97.1 [85.08 to 99.93]

ADVERSE EVENTS:
Time Frame: SAEs and nonserious unsolicited AEs: Day 1 through Day 387; solicited AEs: Day 1 through Day 7 and Day 22 through Day 28
Description: SAEs, nonserious unsolicited AEs, and solicited AEs are reported in this Adverse Events section
Arm/Group | Lowest Dose, Less Adjuvant aH5N1 Vaccine | Low Dose, Less Adjuvant aH5N1 Vaccine | Mid Dose, Less Adjuvant aH5N1 Vaccine | Lowest Dose, Adjuvanted aH5N1 Vaccine | Low Dose, Adjuvanted aH5N1 Vaccine | Mid Dose, Adjuvanted aH5N1 Vaccine
All-Cause Mortality (participants affected / at risk) | 0/69 | 1/72 | 0/70 | 0/70 | 0/69 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/69 | 1/72 | 3/70 | 0/70 | 1/69 | 3/70
Other Adverse Events (participants affected / at risk) | 37/69 | 34/72 | 40/70 | 39/70 | 37/69 | 33/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lowest Dose, Less Adjuvant aH5N1 Vaccine (N=69) | Low Dose, Less Adjuvant aH5N1 Vaccine (N=72) | Mid Dose, Less Adjuvant aH5N1 Vaccine (N=70) | Lowest Dose, Adjuvanted aH5N1 Vaccine (N=70) | Low Dose, Adjuvanted aH5N1 Vaccine (N=69) | Mid Dose, Adjuvanted aH5N1 Vaccine (N=70)
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lowest Dose, Less Adjuvant aH5N1 Vaccine (N=69) | Low Dose, Less Adjuvant aH5N1 Vaccine (N=72) | Mid Dose, Less Adjuvant aH5N1 Vaccine (N=70) | Lowest Dose, Adjuvanted aH5N1 Vaccine (N=70) | Low Dose, Adjuvanted aH5N1 Vaccine (N=69) | Mid Dose, Adjuvanted aH5N1 Vaccine (N=70)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 4 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 12 | 1 | 5 | 5
Injection site erythema (General disorders) | 4 | 5 | 7 | 5 | 5 | 4
Injection site induration (General disorders) | 3 | 3 | 4 | 5 | 5 | 4
Injection site tenderness or pain (General disorders) | 21 | 12 | 17 | 17 | 19 | 17
Change of eating habits (Metabolism and nutrition disorders) | 7 | 8 | 3 | 4 | 6 | 4
Diarrhea (Gastrointestinal disorders) | 10 | 12 | 11 | 10 | 6 | 6
Fatigue (General disorders) | 1 | 2 | 4 | 4 | 6 | 3
Fever (≥38.0°C) (General disorders) | 8 | 9 | 7 | 7 | 2 | 6
Headache (Nervous system disorders) | 3 | 2 | 2 | 3 | 3 | 4
Irritability (Psychiatric disorders) | 8 | 9 | 4 | 6 | 10 | 4
Sleepiness (Nervous system disorders) | 9 | 7 | 5 | 6 | 8 | 3
Vomiting (Gastrointestinal disorders) | 3 | 5 | 5 | 6 | 4 | 1
Other solicited AE (General disorders) | 6 | 6 | 5 | 3 | 4 | 5 — Analgesic/antipyretic use for prevention of pain/fever
Other solicited AE (General disorders) | 7 | 7 | 5 | 3 | 4 | 7 — Analgesic/antipyretic use for treatment of pain/fever

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04669691/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT04669691/SAP_001.pdf